CLINICAL TRIAL: NCT05580445
Title: A Phase Ib/II, Open-label, Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antineoplastic Activity of CT-707 in Combination With Toripalimab and Gemcitabine in Advanced Pancreatic Cancer
Brief Title: Safety, Pharmacokinetics and Efficacy of CT-707, Toripalimab and Gemcitabine in Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-707-1
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Advanced Pancreatic Cancer
Keywords: CT-707, Focal Adhesion Kinase, Advanced Pancreatic Cancer
MeSH Terms: interventions — conteltinib; toripalimab; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation and dose-expansion (Experimental): Dose-escalation study is designed to determine the dose-limiting toxicity (DLTs) and recommended phase II dose (RP2D). Dose-expansion study is designed to evaluate the antitumor activity of CT-707 in combination with toripalimab and gemcitabine in patients with advanced pancreatic cancer.
  Interventions: Drug: CT-707; Drug: Toripalimab; Drug: Gemcitabine

INTERVENTIONS:
Drug: CT-707 — Focal Adhesion Kinase (FAK) inhibitor
  Other Names: CT-707 granules
Drug: Toripalimab — Programmed Death 1(PD-1) antibody
  Other Names: Toripalimab injection
Drug: Gemcitabine — nucleoside inhibitor
  Other Names: GEMZAR

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics and antineoplastic activity of CT-707 in combination with toripalimab and gemcitabine in patients with advanced pancreatic cancer

DETAILED DESCRIPTION:
This is a phase Ib/II, open-label, dose-escalation and dose-expansion study to evaluate the safety, tolerability, pharmacokinetics and antineoplastic activity of CT-707 in combination with toripalimab and gemcitabine in patients with advanced pancreatic cancer.The study consists of two parts, dose-escalation part and dose-expansion part. Both parts will enroll patients with advanced pancreatic cancer. Dose-escalation study is designed to determine the dose-limiting toxicity (DLTs) and recommended phase II dose (RP2D), and to characterize the safety, tolerability, and pharmacokinetics (PK) profile of CT-707 in combination with toripalimab and gemcitabine. Dose-expansion study phase is designed to evaluate the antitumor activity (objective response rate, progression-free survival, overall survival) of CT-707 in combination with toripalimab and gemcitabine in patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in this study, patients must fulfil the following criteria:

  1. Male or female (age of 18~75 years old).
  2. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  3. Patients must have a life expectancy of ≥ 3 months.
  4. Patients must have histologically or cytologically confirmed advanced pancreatic adenocarcinoma or poorly differentiated pancreatic carcinoma that is metastatic to distant sites.
  5. Patients are required to have measurable disease (RECIST v1.1), defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral CT scan.
  6. Patients must have adequate organ and marrow function as defined below:

     Blood routine: Absolute neutrophil count (ANC) ≥ 1.5×10^9/L; Platelet count (PLT) ≥ 100×10^9/L; Hemoglobin (HGB) ≥ 90 g/L.

     Liver function: Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 times upper limit of normal (ULN), total bilirubin (TBIL) ≤ 1.5 times ULN in patients without liver metastases; AST and ALT ≤ 5 times ULN, TBIL ≤3 times ULN in patients with liver metastases.

     Renal function: Serum creatinine (Scr) ≤1.5 times ULN or creatinine clearance ≥60 mL/min/1.73 m2.

     Coagulation function: Activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; International Normalized ratio (INR) ≤ 1.5 times ULN.
  7. Patients must have recovered from any acute adverse events (except alopecia and peripheral neurotoxicity ≤ Grade 2).
  8. Patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial and for 6 months after the trial; female participants must have a negative serum pregnancy test within 7 days prior to treatment.

Exclusion Criteria:

* Patients must not enroll in this study if any of the following exclusion criteria are fulfilled:

  1. Patients who have received chemotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor therapy within 4 weeks prior to the first use of the study drug.
  2. Patients who have received clinical investigational drug or treatment within 4 weeks prior to the first use of the study drug.
  3. Patients who have received major surgery within 4 weeks or had minor surgery within 2 weeks before the first dose of administration.
  4. Patients who have previously received FAK inhibitor or programmed cell death protein 1/programmed cell death ligand 1 (PD-1/L1) antibody and cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) antibody are not eligible.
  5. Patients receiving any medications or substances that are known to be moderate to strong inhibitors or inducers of CYP3A4 and which cannot be discontinued at least 1 week prior to the first dose of administration .
  6. Patients who have active central nervous system (CNS)or leptomeningeal metastasis. However, participants who are asymptomatic, clinically stable, and did not require steroid therapy at least 4 weeks before the first dose of study treatment are eligible.
  7. Patients who have cardiovascular and cerebrovascular diseases currently or within the last 6 months, including but not limited to:

     I. Myocardial infarction; II. Unstable Angina pectoris; III. Cerebrovascular accident; IV. Other acute uncontrolled heart disease; Mean resting corrected QTc interval using the Fridericia formula (QTcF) > 470 msec/female and > 450 msec/male; Severe arrhythmias or abnormal cardiac conduction, such as ventricular arrhythmias requiring clinical intervention, degree ii-iii atrioventricular block, etc; Various factors that may increase the risk of QTc prolongation or arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, a family history of a first-degree relative with long QT syndrome or sudden unexplained death before the age of 40, receiving any medication with known QT prolongation; Left ventricular ejection fraction (LVEF) < 40 % within 4 weeks prior to the first use of the study drug; Hypertension remains uncontrolled after aggressive antihypertensive therapy. Uncontrolled hypertension was defined as systolic blood pressure > 185 mmHg and/or diastolic blood pressure > 110 mmHg measured on 3 repetitions at least 10 minutes apart.
  8. Patients suffering from conditions which are likely to adversely affect gastrointestinal motility (ulcerative disease, uncontrollable nausea, vomiting, diarrhea, or poor absorption syndrome).
  9. Any evidence of severe or uncontrolled systemic disease, active infection or active bleeding diatheses, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
  10. Patients have uncontrolled pleural, pericardial or abdominal effusion requiring drainage excluding those staying stable for at least two weeks after drainage.
  11. Patients have active autoimmune disease that requires systemic treatment (immunomodulatory drugs, corticosteroids, or immunomodulatory drugs) in the past 2 years.
  12. Patients with severely impaired lung functions such as pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia and drug-associated pneumonia.
  13. Patients have allergic reactions to any component of CT-707, toripalimab and gemcitabine, or with history of severe allergic reactions to other monoclonal antibodies or gemcitabine.
  14. Female patients who are pregnant or breast-feeding, or male or female patients of reproductive potential who are not employing an effective method of birth control.
  15. Patients with mental disorder, alcohol and/or drug dependence.
  16. The investigator considers that the subject has a history of serious systemic diseases or other reasons and is not suitable or not willing to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-08-11 (Estimated); Study Completion 2024-08-11 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of CT-707 in combination with toripalimab and gemcitabine | Up to 24 months
  The RP2D will be determined from the maximum tolerated dose (MTD) found in the dose-escalation cohort. The MTD is determined as the dose at which no more than one patient (out of six) experiences any drug-related toxicity (DLT)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | Up to 24 months
  Characterization of the safety and tolerability as determined by changes in laboratory values and electrocardiograms
Pharmacokinetics (Cmax) for CT-707 | Cycle 1 (each cycle is 21 days)
  Defined as maximum observed plasma concentration
Pharmacokinetics (Tmax) for CT-707 | Cycle 1 (each cycle is 21 days)
  Defined as time to maximum plasma concentration
Pharmacokinetics (AUC0-t) for CT-707 | Cycle 1 (each cycle is 21 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Pharmacokinetics (t½) for CT-707 | Cycle 1 (each cycle is 21 days)
  Defined as the apparent plasma terminal phase disposition half-life
Overall response rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary measure of anti-tumor activity of CT-707 in combination with toripalimab and gemcitabine
Progression free survival (PFS) according to RECIST v1.1 criteria | Up to 24 months
  Preliminary measure of anti-tumor activity of CT-707 in combination with toripalimab and gemcitabine
Disease control rate (DCR) according to RECIST v1.1 | Up to 24 months
  Preliminary measure of anti-tumor activity of CT-707 in combination with toripalimab and gemcitabine

OTHER OUTCOMES:
Predictive biomarkers for response to the combination of CT-707, toripalimab and gemcitabine | Up to 24 months
  To assess putative predictive biomarkers such as PD-L1 and p-FAK

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China